CLINICAL TRIAL: NCT01212705
Title: Effect of Adaptive Servoventilation on Cardiac Function, Exercise Tolerance and Quality of Life in Patients With Chronic Heart Failure and Cheyne-Stokes Respiration
Brief Title: Effect of Adaptive Servoventilation on Cardiac Function in Chronic Heart Failure and Cheyne-Stokes Respiration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Other Study IDs: BW2126/10
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Heart Failure; Central Sleep Apnea; Cheyne-Stokes Respiration
MeSH Terms: conditions — Sleep Apnea, Central; Cheyne-Stokes Respiration

ARMS (1):
- ASV (Experimental)
  Interventions: Device: Adaptive servoventilation

INTERVENTIONS:
Device: Adaptive servoventilation — Background expiratory positive airway pressure with some inspiratory pressure support when needed

SUMMARY:
Sleep disordered breathing is common in patients with chronic heart failure. Adaptive servoventilation is a novel method of treatment central sleep apnoea, especially associated with Cheyne-Stokes-respiration. The aim of the study is to investigate effect of adaptive servoventilation on cardiac function, exercise tolerance and quality of life in patients with chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure with ejection fraction ≤45%
* optimal medical treatment for at least 1 month
* clinical diagnosis of Cheyne-Stokes respiration

Exclusion Criteria:

* unstable heart failure
* stroke
* transient ischemic attack in last 6 months
* pacemaker, cardioverter-defibrillator or resynchronization device implanted less than 6 months before study entrance
* severe chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kazimierczak, Principal Investigator — Military Institute of Medicine
Locations (1):
- Military Institute of Medicine, Warsaw, Szaserow 128, Poland